CLINICAL TRIAL: NCT00485342
Title: Multicentric, Controlled and Randomised Open Clinical Trial Investigating the Efficacy and Safety of Dose Adaptation of Ribavirin Using Pharmacologic Measures of Ribavirin Exposition During Combination Peginterferon Alfa-2 and Ribavirin Treatment in Naive Patients With Chronic Hepatitis C of Genotype 1 on a First Combination Therapy
Brief Title: RIBAJUSTE Clinical Trial Investigating the Efficacy and Safety of Dose Adaptation of Ribavirin
Acronym: RIBAJUSTE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-400
Record Dates: First submitted 2007-06-08; First posted 2007-06-12 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C,Genotype1,Naïf,bitherapy,Ribavirin adaptation,ribavirin AUC
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard dose (No Intervention): the "reference" strategy : Peg-interferon alpha 2a (180 µg/week) and ribavine (1000 mg/day if weight < 75 kg and 1200 mg/day if weight ≥ 75 kg)
  Interventions: Drug: Peg-interferon alpha 2a and ribavin
- adjusted dose (Experimental): individual dose adjustment of ribavirin dose at D7, based on ribavirin abbreviated AUC-0-4H , estimated itself by two independent methods: multiple linear regression and bayesien estimation based on three ribavirin concentration measurements obtained at 0.5H, 1H, 2H after the first intake of 600 mg at D0.
  Interventions: Drug: ribavirin with adaptation dose

INTERVENTIONS:
Drug: Peg-interferon alpha 2a and ribavin — Date of ribavirin AUC : Day 0 (beginning of treatment) Bitherapy : Peg-interferon alpha 2a (180 µg/week) with ribavirin (1000 mg/day if weight < 75 kg and 1200 mg/day if weight ≥ 75 kg).
  Duration of treatment : 48 weeks Duration of study for patients : 72 weeks
  Arms: standard dose
Drug: ribavirin with adaptation dose — Date of ribavirin AUC : Day 0 (beginning of treatment) Bitherapy : Peg-interferon alpha 2a (180 µg/week) with ribavirin (dose adaptation) Dose adaptation : Day 7, dependant of result of AUC Ribavirin dose increments : 200 mg, 400 mg or 600 mg with a maximum of 50% of the initial dose (600 mg) applied every 4 days up to the adjusted dose proposed in order to reach the targeted AUC.
  The maximum daily dose will not exceed 3600 mg Duration of treatment : 48 weeks Duration of study for patients : 72 weeks
  Arms: adjusted dose

SUMMARY:
The aim of this study is to compare two therapeutical strategies concerning the combination therapy (peginterferon alfa-2a and ribavirin) in naïve patients with chronic hepatitis C of genotype 1. "Reference" strategy corresponding to standards of care recommended by the French consensus conference versus "Test" strategy corresponding to adaptation strategy of ribavirin dose during the first week according to AUC (area under the curve) of ribavirin plasmatic concentration after the first intake (Day 0) of 600 mg

ELIGIBILITY:
Inclusion Criteria:

* 65 years >Age >= 18 years
* Chronic hepatitis C documented by PCR performed within 3 months and at liver biopsy within 18 months or with serum markers of fibrosis performed within 3 months before inclusion or FibroScan performed
* Naive patients for who the physician decided to initiate a combination treatment of chronic hepatitis C with pegylated interferon alfa-2a plus ribavirine
* Genotype VHC-1
* Compensated liver disease (Child-Pugh <=6)
* Negative HBsAg test and HIV-RNA test
* Negative pregnancy test at baseline in women in age of procreation and efficient contraception all along the treatment period, and up to 7 months after discontinuation for women and men
* Signed consent form
* Patient with a social cover

Exclusion Criteria:

* Non HCV liver disease
* Non-1 HCV genotype
* Organ transplant whatever the organ
* Clinical or radiological evidence of liver carcinoma
* Severe psychiatric disorder
* Non compensated thyroid dysfunction
* Woman pregnant or breast-feeding
* Recent history of epilepsy (less than 6 months)
* Absolute contraindications to one of the drug of combination therapy
* Biological abnormalities at pre-treatment check-up, such as:

Neutropenia (<1500/mm³); Haemoglobinemia (<13 g/dL for men et <12 g/dL for women); Thrombopenia (<90 000/mm³);

* Kidney failure (creatinine clearance>70 ml/min)
* Hypersensitivity to epoetin or one of its excipients
* Treatment by epoetin within 2 months prior inclusion
* Chronic cardiac failure (grade III or IV - NYHA classification)
* High blood pressure unwell-controlled (SBP > 180 mmHg during inclusion in spite of hypertension treatment)
* Previous history or risk of venous thrombosis
* Major surgery within the previous 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2006-04; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Inter-group comparison of sustained virological response rates as defined by the proportion of subjects with a negative PCR HCV-RNA test at Week 72 | 72 weeks

SECONDARY OUTCOMES:
Efficacy endpoints | 72 weeks
  To compare the virological response rate between the two groups: Rapid Virological Response (RVR) at W4, Early Virological Response (EVR) at W12, Virological Response at W24, and End-Of-Treatment response (EOT) at W48 ; To determine the relapse rate (between W48 and W72) and to determine the proportion of patients reaching the target trough ribavirin concentration of 2 mg/L at W4 or W8 after ribavirin dose adjustment in the first 7 days of treatment.
safety endpoints | 72 weeks
  To investigate the clinical and biological tolerability in patients with dose-adjusted ribavirin compared to those with standard ribavirin doses, the proportion of patients needing EPO co-prescription due to secondary anemia in each group, to estimate the rate of treatment discontinuation due to serious or other relevant adverse events in each group and to determine the proportion of subjects reaching ribavirin trough plasma concentrations considered as "toxic" (> 3.5 mg/L) at W4 and W8, in each arm.
Economic endpoints | 72 weeks
  Comparaison of the "test" and "standard" strategies by a medico-economic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christian Trépo, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Marianne Maynard, Lyon, France